CLINICAL TRIAL: NCT04110301
Title: A Multi-center, Open Label, Phase 1b/2 Study to Study the Efficacy and Safety of MIL62 Plus Lenalidomide in Subjects With Relapsed/Refractory Follicular Lymphoma or Marginal Zone Lymphoma
Brief Title: MIL62 Plus Lenalidomide for Patients With Relapsed/Refractory Indolent Non-Hodgkin's Lymphoma (FL and MZL)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Beijing Mabworks Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MIL62-CT02
Record Dates: First submitted 2019-09-27; First posted 2019-10-01 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-10

CONDITIONS: Follicular Lymphoma and Marginal Zone Lymphoma
Keywords: CD20 ,Follicular Lymphoma,Marginal Zone Lymphoma,MIL62
MeSH Terms: conditions — Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MIL62 + Lenalidomide (Experimental): MIL62 plus Lenalidomide
  Interventions: Drug: Recombinant Humanized Monoclonal Antibody MIL62 Injection; Drug: Lenalidomide

INTERVENTIONS:
Drug: Recombinant Humanized Monoclonal Antibody MIL62 Injection — 1000mg /dose for 12 cycles(28 days) and a total of 11 doses :the first Cycle(Day1,Day15), the 2nd-8th Cycles(Day 1 every cycle);the 9th-12nd Cycles (One dose every two cycles).
  Other Names: MIL62
Drug: Lenalidomide — Dose on days 2-22 every 28 days x 12 cycles: the starting dose is 10-mg ; Adjusted dose according to the tumor response or toxicity reaction
  Other Names: Revlimid

SUMMARY:
This phase 1b/2 trial studies the safety and best dose of lenalidomide when given together with MIL62 and how well this combination works in treating patients with Relapsed/Refractory low-grade Follicular Lymphoma(FL) and Marginal Zone Lymphoma(MZL). Giving MIL62 plus lenalidomide may work better in indolent Non-Hodgkin Lymphoma(NHL).

DETAILED DESCRIPTION:
The Aim of this phase 1b/2 trial (MIL62 Plus Lenalidomide) is to find the safety and best dose of lenalidomide when given together with MIL62 and how well this combination works in treating patients with Relapsed/Refractory low-grade Follicular Lymphoma(FL) and Marginal Zone Lymphoma(MZL). Giving MIL62 plus lenalidomide may work better in indolent Non-Hodgkin Lymphoma(NHL).

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients, >=18 years of age;
2. Patients with either histologically documented CD20-positive MZL or FL, WHO grade 1, 2 or 3a
3. Evidence of progression or lack of response following at least 1 prior treatment
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2
5. At least one bi-dimensionally measurable nodal or tumor lesion defined by CT scan as: greatest transverse diameter > 1.5 cm and a short axis ≥ 10mm
6. Adequate hematologic function (unless abnormalities are related to NHL)
7. Life expectancy >6 months
8. Able and willing to provide written informed consent and to comply with the study protocol

Exclusion Criteria:

1. Evidence ongoing transformation into aggressive NHL
2. Central nervous system lymphoma
3. Patients with progressive multifocalleukoencephalopathy (PML)
4. Prior use of any antibody therapy(except for Rituximab ) within 3 months of study start
5. Prior use of any anti-cancer vaccine
6. Prior administration of radiotherapy 42 days prior to study entry
7. Prior administration of chemotherapy 28 days prior to study entry
8. History of prior malignancy within the last 3 years, with the exception of curatively treated basal or squamous cell carcinoma of the skin and low-grade in situ carcinoma of the cervix
9. History of severe allergic or anaphylactic reactions to monoclonal antibody therapy
10. Known hypersensitivity to thalidomide or lenalidomide
11. Regular treatment with corticosteroids prior to the start of cycle 1, unless administered for indications other than NHL at a dose equivalent to < 20 mg/day prednisone
12. Any serious active disease or co-morbid medical condition (such as New York Heart Association Class II or IV cardiac disease, severe arrhythmia, myocardial infarction within the last 6 months, unstable arrhythmias, or unstable angina) or pulmonary disease (including obstructive pulmonary disease and history of bronchospasm or other according to investigator's decision)
13. Infection with human immunodeficiency virus (HIV), hepatitis B or hepatitis C(including HBsAg,HBcAb positive with abnormal HBV DAN or HCV RNA )
14. Pregnant or lactating females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2019-11-28 (Actual); Primary Completion 2024-01-09 (Actual); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With an Objective Response of Complete Response | Baseline to 1 month after the last dose of last patient
  Percentage of Participants With an Objective Response of Complete Response

SECONDARY OUTCOMES:
Kaplan-Meier Estimate of Duration of Response | Baseline to 1 month after the last dose of last patient
  Kaplan-Meier Estimate of Duration of Response
Percentage of Participants With Disease Control | Baseline to 1 month after the last dose of last patient
  Percentage of Participants With Disease Control
Participants With 1 Year Progression Free Survival | Baseline to 1 month after the last dose of last patient
  Participants With 1 Year Progression Free Survival
Number of Participants With Treatment Emergent Adverse Events | up to the 1 month the last dose of last subject
  Number of Participants With Treatment Emergent Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Yuankai Shi, MD, Principal Investigator — Cancer Institute&Hospital, Chinese Academy of Medical Sciences,Beijing
Locations (1):
- Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, China

REFERENCES:
- [Derived] Shi Y, Zhou K, Zhou H, Qin Y, Jing H, Xiang Y, Wang Z, Wang Z, Zang A, Bai O, Li Z, Zhang H, Song Y, Liang J, Wei M. Efficacy and safety of MIL62, a novel glycoengineered type Ⅱ anti-CD20 monoclonal antibody, combined with lenalidomide in patients with relapsed/refractory follicular lymphoma or marginal zone lymphoma: a multicentre, single-arm, phase 1b/2 trial. EClinicalMedicine. 2024 Jun 20;73:102702. doi: 10.1016/j.eclinm.2024.102702. eCollection 2024 Jul. PMID 39007066